CLINICAL TRIAL: NCT06672133
Title: Adebrelimab Combined with Chemotherapy and Thoracic Radiotherapy for First-line Treatment of ES-SCLC: a Randomized Controlled Phase III Clinical Study
Brief Title: Adebrelimab Combined with Chemotherapy and Thoracic Radiotherapy for First-line Treatment of ES-SCLC
Acronym: RALLY
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jinming Yu (Other)
Responsible Party: Sponsor-Investigator, Jinming Yu, President of Shandong Cancer Hospital，Academician of Chinese Academy of Engineering, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-SCLC-III-023
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma
Keywords: adebrelimab; radiotherapy; ES-SCLC
MeSH Terms: interventions — Radiotherapy; Radiation

STUDY DESIGN:
Intervention Model Description: Subjects who had SD/PR/CR assessed after induction immunotherapy were randomized 1:1 with PFS and OS set as co-primary endpoints for this study.
  The HR of mOS in the maintenance phase was conservatively estimated to be meaningful in the adalimumab combined with thoracic radiotherapy group compared with the adalimumab group, with a significance level α of 0.05 (2-sided), and no less than 80% OS events would be observed (1-β difference between the 375 groups).
  A total of 471 subjects are required to be enrolled. Considering a dropout rate of 10%, 524 subjects were required. In summary, a total of at least 524 subjects were required to be enrolled in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm Combined Radiotherapy (Experimental): After randomization，patients receive adebrelimab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo radiation therapy QD on days 1-5 during weeks 1-5 only.
  Patients undergo CT, MRI or PET/CT scan,throughout the trial. Patients also undergo blood and tissue collection throughout the trial.
  Interventions: Drug: Adebrelimab; Radiation: Radiation Therapy
- Arm Non-radiotherapy (Active Comparator): After randomization，patients receive adebrelimab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Patients undergo CT, MRI or PET/CT scan,throughout the trial. Patients also undergo blood and tissue collection throughout the trial.
  Interventions: Drug: Adebrelimab

INTERVENTIONS:
Drug: Adebrelimab — Given：IV
  Other Names: SHR-1316
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: RT; Radiotherapy; Consolidation radiotherapy; Irradiation
  Arms: Arm Combined Radiotherapy

SUMMARY:
This phase III trial compares the effect of adding radiation therapy to the usual maintenance therapy with adebrelimab versus adebrelimab alone in patients who have already received debrelimab plus chemotherapy for the treatment of extensive stage small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I.To compare investigator-assessed progression free survival (PFS) between adebrelimab plus radiotherapy and adebrelimab alone.

II.To compare overall survival (OS) between adebrelimab plus radiotherapy and adebrelimab alone.

SECONDARY OBJECTIVES:

I.To assess the ORR (objective response rate)、DoR (Duration of response) 、DCR(Disease control rate) toxicity between the adebrelimab plus radiotherapy arm and the adebrelimab arm.

II.To assess six months and one-year PFS rate、one-year and two-year OS rate between the adebrelimab plus radiotherapy arm and the adebrelimab arm.

III.To assess the safety and tolerability.

EXPLORATORY OBJECTIVE:

I.To detect biomarkers associated with efficacy OUTLINE: Patients are randomized to 1 of 2 arms. ARM I: Patients receive adebrelimab IV over 30 minutes. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo radiation therapy once daily (QD) on days 1-5 during weeks 1-5 only.

ARM II: Patients receive adebrelimab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients undergo computed tomography (CT)、magnetic resonance imaging (MRI) or positron emission tomography and computed tomography (PET/CT) scan, throughout the trial. Patients also undergo blood and tissue collection throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, male or female;
2. Histologically or cytologically confirmed extensive stage small cell lung cancer (according to the Veterans Lung Administration Lung Study Group, VALG stage);
3. ECOG performance status score 0 ~ 1;
4. No prior line of systemic therapy for ES-SCLC;
5. Liver metastases ≤ 3 at diagnosis;
6. Patients without previous brain metastases or treated asymptomatic CNS metastases,
7. Expected survival ≥ 12 weeks;
8. At least one measurable target lesion (according to RECISTv1.1 criteria) on imaging assessment (CT or MRI) within 4 weeks prior to enrollment;
9. The function of vital organs meets the requirements;
10. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose and must agree to use effective contraception during the trial and 2 months after the last dose of adalimumab or 6 months after the chemotherapy agent, whichever is longer;
11. Patients voluntarily join this study, sign informed consent, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Histologically or cytologically determined as a mixed pathological type with components such as non-small cell lung cancer;
2. Active or untreated CNS metastases detected by computed tomography (CT) or magnetic resonance imaging (MRI) during the screening period and previous imaging assessments;
3. Spinal cord compression that is not relieved by surgery and/or radiotherapy;
4. Clinically symptomatic third space effusion requiring repeated drainage within 2 weeks, such as pericardial effusion, pleural effusion, and abdominal effusion that are still uncontrollable by pumping or other treatments;
5. Complicated with other malignant tumors ≤ 5 years before the first dose, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical resection, and ductal carcinoma in situ after radical resection (hormone therapy for non-metastatic prostate cancer or breast cancer is allowed);
6. Patients with active, known, or suspected autoimmune disease. Patients with type 1 diabetes treated with stable doses of insulin, hypothyroidism requiring hormone replacement therapy only, and skin diseases (e.g., eczema, vitiligo, or psoriasis) not requiring systemic therapy and not exacerbated within the year before the screening period were excluded;
7. Patients diagnosed with immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy not directly related to tumor therapy within 7 days before the first dose of study drug; physiological doses of glucocorticoids (prednisone ≤ 10 mg/day or equivalent) are allowed;
8. HBsAg positive and HBV DNA copy number greater than the upper limit of normal (1000 copies/ml or 500 IU/ml), or HCV positive (HCV RNA or HCV Ab detection suggests acute and chronic infection); known HIV positive history or known acquired immunodeficiency syndrome (AIDS);
9. A history of idiopathic pulmonary fibrosis, interstitial pneumonia, tissue pneumonia (such as occlusive vasculitis), drug-induced pneumonia, radiation pneumonitis requiring steroid therapy or clinically symptomatic active pneumonia; or other severe lung disease that seriously affects lung function;
10. Patients with active pulmonary tuberculosis (TB) or history of active pulmonary tuberculosis infection ≤ 48 weeks before screening, regardless of treatment;
11. Presence of severe infection at randomization, including but not limited to infectious complications requiring hospitalization, bacteremia, severe pneumonia, etc.;
12. Major surgery within 28 days prior to randomization, or planned major surgery during the study period;
13. Use of live attenuated vaccines within 28 days prior to randomization, or anticipated need for live attenuated vaccines during the study;
14. Cardiac function and disease which is considered clinically significant by the investigator;
15. Patients who have previously received allogeneic bone marrow transplantation or solid organ transplantation;
16. Known hypersensitivity to the study drug or excipients, known serious allergic reactions to any monoclonal antibody; history of allergy to carboplatin/cisplatin or etoposide;
17. Received any other investigational drug or participated in another interventional clinical study within 4 weeks before signing the ICF;
18. Known mental illness, alcoholism, inability to quit smoking, drug abuse or drug abuse;
19. Pregnant or lactating women; as judged by the investigator, the patient has other factors that may cause forced halfway termination of this study, such as non-compliance with the protocol, other serious diseases (including mental illness) requiring concomitant treatment, severe laboratory abnormalities, accompanied by family or social factors, which may affect the safety of patients, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to approximately 36 months
OS | Up to approximately 36 months

SECONDARY OUTCOMES:
ORR | Up to approximately 36 months
DoR | Up to approximately 36 months
DCR | Up to approximately 36 months
6m and 1-year PFS rate | 6 Months and 12 Months
1- and 2-year OS rates | 1 year and 2 years
Adverse events | Up to approximately 36 months
  Safety, incidence and severity of adverse events (AEs) and serious adverse events (SAEs) per CTCAE 5.0 criteria

OTHER OUTCOMES:
To detect biomarkers associated with efficacy | Up to approximately 36 months

IPD SHARING:
Plan to Share IPD: No